CLINICAL TRIAL: NCT03782532
Title: A Randomized, Double Blind, Placebo-controlled, Parallel-group Phase 3 Study to Evaluate the Efficacy and Safety of Dupilumab in Patients With Persistent Asthma
Brief Title: Efficacy and Safety Study of Dupilumab in Patients With Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC13995; U1111-1175-0772 (Other: UTN); 2022-002375-11 (EudraCT Number)
Record Dates: First submitted 2018-12-05; First posted 2018-12-20 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): For patients without oral corticosteroids (OCS) maintenance therapy, dose 1 of dupilumab administered once in 2 weeks (q2w) with loading dose of dupilumab, two times dose 1; for patients on OCS maintenance therapy, the dose will be dupilumab dose 2 q2w with loading dose 2 times dose 2
  Interventions: Drug: Dupilumab SAR231893; Drug: Asthma Controller Therapies (include prednisone/prednisolone); Drug: Asthma Reliever Therapies
- Placebo for dupilumab (Placebo Comparator): For patients without OCS maintenance therapy, the patients will take placebo matching to dupilumab dose 1 q2w with loading dose; for patients on OCS maintenance therapy, the patients will take placebo matching to dupilumab dose 2 q2w with loading dose
  Interventions: Drug: Placebo; Drug: Asthma Controller Therapies (include prednisone/prednisolone); Drug: Asthma Reliever Therapies

INTERVENTIONS:
Drug: Dupilumab SAR231893 — Pharmaceutical form: Solution
  Route of administration: Subcutaneous
  Arms: Dupilumab
Drug: Placebo — Pharmaceutical form: Solution
  Route of administration: Subcutaneous
  Arms: Placebo for dupilumab
Drug: Asthma Controller Therapies (include prednisone/prednisolone) — Pharmaceutical form: Aerosol, capsules, tablets, oral solution
  Route of administration: Inhalation, oral
Drug: Asthma Reliever Therapies — Pharmaceutical form: Nebulized, aerosol
  Route of administration: Inhaled

SUMMARY:
Primary Objective:

To evaluate the efficacy of dupilumab in patients with persistent asthma

Secondary Objectives:

* To evaluate the safety and tolerability of dupilumab
* To evaluate the effect of dupilumab on improving patient reported outcomes including health related quality of life
* To evaluate dupilumab systemic exposure and immunogenicity

DETAILED DESCRIPTION:
The total duration of study per patient is approximately 40 weeks, including 3 to 5 weeks of screening period, 24 weeks of treatment period and 12 weeks of post-treatment period.

ELIGIBILITY:
Inclusion criteria :

* Adults and adolescent patients (≥12 years of age) with a physician diagnosis of asthma for ≥12 months, based on the Global Initiative for Asthma 2017 Guidelines and the following criteria:
* Patients requiring a third controller for their asthma will be considered eligible for this study, and it should also be used for at least 3 months with a stable dose ≥1 month prior to the screening visit (Visit 1).
* Patients requiring maintenance oral corticosteroids (OCS) with a stable dose ≤10 mg/day prednisone or equivalent will be allowed; OCS should be used for at least 3 months with a stable dose ≥1 month prior to the screening visit (Visit 1).
* Pre-bronchodilator FEV1 ≤ 80% of predicted normal for adults and ≤90% of predicted normal for adolescents at the screening visit and the randomization visit (Visits 1 and 2), prior to randomization.
* Asthma Control Questionnaire 5-question version (ACQ-5) score ≥1.5 at the screening visit and the randomization visit (Visits 1 and 2), prior to randomization.
* For patients not requiring maintenance OCS, screening blood eosinophil count ≥150 cells/μL or Fractional Exhaled Nitric Oxide (FENO) ≥25 parts per billion (ppb); for patients requiring maintenance OCS, there is no minimum requirement for blood eosinophil count and FENO level.

Exclusion criteria:

* Patients <12 years of age or the minimum legal age for adolescents in the country of the investigative site, whichever is higher (for those countries where local regulations permit enrollment of adults only, patient recruitment will be restricted to those who are ≥18 years of age).
* Weight is less than 30 kg at the screening visit (Visit 1) or the randomization visit (Visit 2).
* Chronic obstructive pulmonary disease or other lung diseases (eg, idiopathic pulmonary fibrosis) which may impair lung function.
* A patient who experiences a severe asthma exacerbation (defined as deterioration of asthma that results in emergency treatment, hospitalization due to asthma, treatment with systemic steroids, or treatment with systemic steroid at least twice the previous dose for patients on OCS maintenance) at any time from 1 month prior to the screening visit (Visit 1) up to and including the randomization visit (Visit 2).
* Evidence of lung disease(s) other than asthma, either clinical or imaging evidence (eg, chest X-ray, computed tomography, and magnetic resonance imaging) within 3 months prior to the screening visit (Visit 1) as per local standard of care.
* Current smoker or cessation of smoking within 6 months prior to the screening visit (Visit 1).
* Previous smoker with a smoking history >10 pack-years.
* Comorbid disease that might interfere with the evaluation of investigational medicinal product (IMP).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
Change in pre-bronchodilator forced expiratory volume (FEV1) | Baseline to Week 12
  Absolute change from baseline in pre-bronchodilator FEV1 at Week 12

SECONDARY OUTCOMES:
Annualized rate of severe exacerbation events | During the 24-week placebo-controlled treatment period
  Annualized rate of severe exacerbation events during the 24-week placebo-controlled treatment period
Percent change from baseline in pre-bronchodilator FEV1 | Baseline to Week 12
  Percent change from baseline in pre-bronchodilator FEV1 at Week 12
Annualized rate of loss of asthma control (LOAC) event | During the 24-week placebo-controlled treatment period
  Annualized rate of LOAC event during the 24-week placebo-controlled treatment period
Annualized rate of severe exacerbation events resulting in hospitalization or emergency room visit | During the 24-week placebo-controlled treatment period
  Annualized rate of severe exacerbation events resulting in hospitalization or emergency room visit during the 24-week placebo-controlled treatment period
Time to first severe exacerbation event | During the 24-week placebo-controlled treatment period
  Time to first severe exacerbation event during the 24-week placebo-controlled treatment period
Time to first LOAC | During the 24-week placebo-controlled treatment period
  Time to first LOAC during the 24-week placebo-controlled treatment period
Change from baseline in Asthma Control Questionnaire (ACQ)-5 score | Baseline to Week 24
  Change from baseline in ACQ-5 score at Week 24
Change from baseline in ACQ-7 score | Baseline to Week 24
  Change from baseline in ACQ-7 score at Week 24
Morning/evening asthma symptom score (e-diary) | Baseline to Week 24
  Change from baseline at Week 24 in morning/evening asthma symptom score (e-diary)
Nocturnal awakenings (e-diary) | Baseline to week 24
  Change from baseline at Week 24 in nocturnal awakenings (e-diary)
Use of daily puffs of rescue medication | Baseline to Week 24
  Change from baseline at Week 24 in use of daily puffs of rescue medication
Change from baseline in Asthma Quality of Life Questionnaire (AQLQ) with Standardized Activities (≥12 years) (AQLQ+12) | Baseline to Week 24
  Change from baseline in AQLQ with Standardized Activities (≥12 years) (AQLQ+12) at Week 24
Change from baseline in European Quality of Life Working Group Health Status Measure 5 Dimensions, 5 Levels (EQ-5D-5L) | Baseline to Week 24
  Change from baseline in EQ-5D-5L at Week 24
Assessment of adverse events (AEs) | Baseline to week 36
  Number of participants with adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (67):
- China (54):
  - Investigational Site Number :1560013, Baotou
  - Investigational Site Number :1560016, Beijing
  - Investigational Site Number :1560029, Beijing
  - Investigational Site Number :1560015, Beijing
  - Investigational Site Number :1560056, Beijing
  - Investigational Site Number :1560057, Changchun
  - Investigational Site Number :1560010, Changsha
  - Investigational Site Number :1560030, Chengdu
  - Investigational Site Number :1560053, Chengdu
  - Investigational Site Number :1560025, Chongqing
  - Investigational Site Number :1560004, Guangzhou
  - Investigational Site Number :1560001, Guangzhou
  - Investigational Site Number :1560045, Guangzhou
  - Investigational Site Number :1560032, Guiyang
  - Investigational Site Number :1560019, Hangzhou
  - Investigational Site Number :1560007, Hangzhou
  - Investigational Site Number :1560014, Hangzhou
  - Investigational Site Number :1560026, Hangzhou
  - Investigational Site Number :1560043, Hangzhou
  - Investigational Site Number :1560038, Hefei
  - Investigational Site Number :1560044, Hohhot
  - Investigational Site Number :1560008, Hohhot
  - Investigational Site Number :1560022, Lanzhou
  - Investigational Site Number :1560024, Nanchang
  - Investigational Site Number :1560051, Nanjing
  - Investigational Site Number :1560054, Nanjing
  - Investigational Site Number :1560037, Nanjing
  - Investigational Site Number :1560035, Pingxiang
  - Investigational Site Number :1560050, Shanghai
  - Investigational Site Number :1560049, Shanghai
  - Investigational Site Number :1560005, Shanghai
  - Investigational Site Number :1560011, Shanghai
  - Investigational Site Number :1560017, Shanghai
  - Investigational Site Number :1560006, Shanghai
  - Investigational Site Number :1560002, Shanghai
  - Investigational Site Number :1560018, Shenyang
  - Investigational Site Number :1560036, Shenyang
  - Investigational Site Number :1560012, Shenzhen
  - Investigational Site Number :1560042, Shenzhen
  - Investigational Site Number :1560003, Shijiazhuang
  - Investigational Site Number :1560041, Shijiazhuang
  - Investigational Site Number :1560031, Suzhou
  - Investigational Site Number :1560048, Taiyuan
  - Investigational Site Number :1560020, Tianjin
  - Investigational Site Number :1560033, Ürümqi
  - Investigational Site Number :1560021, Wenzhou
  - Investigational Site Number :1560052, Wuhan
  - Investigational Site Number :1560028, Wuhan
  - Investigational Site Number :1560040, Xi'an
  - Investigational Site Number :1560046, Xiamen
  - Investigational Site Number :1560027, Xiangtan
  - Investigational Site Number :1560023, Xuzhou
  - Investigational Site Number :1560055, Yangzhou
  - Investigational Site Number :1560047, Zhanjiang
- India (13):
  - Investigational Site Number :3560006, Chandigarh
  - Investigational Site Number :3560002, Coimbatore
  - Investigational Site Number :3560013, Hyderabad
  - Investigational Site Number :3560005, Jaipur
  - Investigational Site Number :3560015, Jaipur
  - Investigational Site Number :3560010, Kolkata
  - Investigational Site Number :3560011, Kozhikode
  - Investigational Site Number :3560012, Mohali
  - Investigational Site Number :3560003, Nagpur
  - Investigational Site Number :3560016, Nagpur
  - Investigational Site Number :3560001, New Delhi
  - Investigational Site Number :3560009, Pune
  - Investigational Site Number :3560007, Vellore

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Zhang Q, Zhong N, Dhooria S, Fu X, Fang H, Lin J, Zhu S, Laws E, Wang Y, Li V, Hu CC, Maloney J, Abdulai RM, Robinson LB. Dupilumab Efficacy and Safety in Patients With Persistent Asthma: Asia-Pacific Region. Clin Exp Allergy. 2025 Aug;55(8):691-700. doi: 10.1111/cea.70005. Epub 2025 Feb 23. PMID 39988927
- See also: 2022-002375-11 EudraCT results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2022-002375-11/results